CLINICAL TRIAL: NCT04056572
Title: A Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of TQ-B3139 in Patients With Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC) Previously Treated With Crizotinib.
Brief Title: Study of TQ-B3139 in Subjects With Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC) Previously Treated With Crizotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3139-II-01
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-05

CONDITIONS: ALK-positive NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3139 (Experimental): TQ-B3139 tablet 600mg administered orally, twice daily.
  Interventions: Drug: TQ-B3139

INTERVENTIONS:
Drug: TQ-B3139 — TQ-B3139 is competitive multi-target protein kinase inhibitor of Met/ALK/ROS.

SUMMARY:
To evaluate the efficacy and safety of TQ-B3139 in subjects with ALK-positive non-small cell lung cancer that have demonstrated progression during or after crizotinib treatment whether or not previously treated with cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 and 75 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
3. Life expectancy ≥12 weeks.
4. Histologically or cytologically confirmed diagnosis of advanced or metastatic NSCLC that is ALK-positive.
5. Has progressive disease during or after crizotinib treatment.
6. Has a measurable disease.
7. Adequate organ system function.
8. Understood and signed an informed consent form.

Exclusion Criteria:

1. Diagnosed and/or treated additional malignancy within 5 years prior to randomization.
2. Hypersensitivity to TQ-B3139 capsule.
3. Has received ALK TKIs other than crizotinib.
4. Has received any cancer therapy within 4 weeks or 5 times of t1/2.
5. Has received major surgery within 4 weeks.
6. Has received any radiotherapy or minor surgery within 2 weeks.
7. Acute toxicity ≥ Grade 2 caused by previous cancer therapy.
8. Has active viral, bacterial and fungal infections within 2 weeks.
9. Has serious cardiovascular diseases.
10. Has currently uncontrollable congestive heart failure.
11. Has continuous arrhythmia ≥ Grade 2, any degree of poor controlled atrial fibrillation or QTc interval > 480ms.
12. Has interstitial fibrosis or interstitial lung disease.
13. Brain metastases with symptom or carcinomatous meningitis.
14. Has active hepatitis B or hepatitis C.
15. Has multiple factors affecting oral medication.
16. Breastfeeding or pregnant women.
17. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 36 months
  The percentage of participants with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 36 months
  The time from randomization to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.
Disease control rate (DCR) | up to 36 months
  Calculated as the percentage of participants with best overall response of CR, PR, stable disease (SD) and Non-CR/Non-progressive disease (PD).
Overall survival (OS) | up to 36 months
  Time from date of randomization to date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun-Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan